CLINICAL TRIAL: NCT00294905
Title: Implementation of an Evidence Based Smoking Cessation Strategy (SMOCC) for Patients With COPD in Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment of patients did not reach sufficient numbers
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 945-16-104
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2007-02

CONDITIONS: COPD
Keywords: COPD; smoking cessation; implementation; patient counseling; general practice
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation

INTERVENTIONS:
Behavioral: Implementation of a combined smoking cessation strategy

SUMMARY:
A controlled study demonstrated that a smoking cessation protocol in routine primary care, specifically targeted at patients with COPD (SMOCC), doubled the quit rates. The protocol was tested under optimal trial conditions, but it is unclear if a large-scale implementation strategy is (cost-)effective. Therefore the present study investigates a large scale implementation strategy in a 2-armed community intervention trial. The research question is how (cost-)effective this implementation strategy is compared to usual implementation procedures.

DETAILED DESCRIPTION:
COPD is an increasing cause of death and morbidity and smoking is its primary cause. Professional smoking cessation treatment is very cost-effective and therefore recommended by national guidelines. A controlled study demonstrated that a smoking cessation protocol in routine primary care, specifically targeted at patients with COPD (SMOCC), doubled the quit rates. The incremental cost-effectiveness ratio (ICER) was Euro 1012 showing that the protocol was cost-effective. The protocol was tested under optimal trial conditions, but it is unclear if a large-scale implementation strategy is (cost-)effective. Therefore the present study investigates an implementation strategy in a 2-armed community intervention trial. General practices (N=150, 2700 smoking patients with COPD) will be randomly allocated to the intervention or control condition. In the control condition the usual dissemination strategy of distributing guidelines and subsequent products through the professional channels (journals, postgraduate education) will take place. In the intervention condition a multifaceted implementation strategy wil be executed aimed at support of the general practice team (outreach education by a facilitator, support for detecting smoking patients with COPD, provision of patient education materials, help desk/website, telephone and e-mail reminders). The research question is how (cost-)effective this implementation strategy is compared to usual implementation procedures. Primary outcome measures will be biochemically validated smoking abstinence at 12 and 18 months. Secondary outcome measures will be counseling contacts and counseling behaviour of professionals and cessation attempts of patients. A process analysis and evaluations by patients and professionals are an integral part of the study. A cost-effectiveness analysis taking a health care sector perspective will be performed and will show the expected costs per practice and an incremental cost-effectiveness ratio (ICER). The study will last 34 months, the intervention period will take 18 months per practice.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Smoking
* Age 40 years or over

Exclusion Criteria:

* Under control of lung specialist
* Not Dutch-speaking
* Serious physical of psychiatric comorbidity
* Under 40 years of age

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2006-03; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures will be biochemically validated smoking abstinence at 12 and 18 months

SECONDARY OUTCOMES:
Secondary outcome measures will be counseling contacts and counseling behaviour of professionals and cessation attempts of patients

CONTACTS AND LOCATIONS:
Overall Officials: R. Grol, PhD, Study Director — Centre for Quality of Care Research (WOK), Radboud University Nijmegen Medical Centre
Locations (1):
- Radboud University Nijmegen Medical Centre, Centre for Quality of Care Research (WOK), 117 Kwazo, Postbus 9101, 6500 Hb, Netherlands

REFERENCES:
- [Background] Hilberink SR, Jacobs JE, Bottema BJ, de Vries H, Grol RP. Smoking cessation in patients with COPD in daily general practice (SMOCC): six months' results. Prev Med. 2005 Nov-Dec;41(5-6):822-7. doi: 10.1016/j.ypmed.2005.08.003. Epub 2005 Oct 3. PMID 16203030
- See also: Site of the Centre for Quality of Care Research (WOK) — http://www.wokresearch.nl